CLINICAL TRIAL: NCT03121170
Title: Extracorporeal Shock Wave Therapy in the Treatment of Primary Dysmenorrhea:a Randomized Controlled-placebo Trial
Brief Title: Extracorporeal Shock Wave Therapy in the Treatment of Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruirui Xing (Other)
Responsible Party: Sponsor-Investigator, Ruirui Xing, Principal Investigator, Master, Xuhui Central Hospital, Shanghai
Organization: Xuhui Central Hospital, Shanghai (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XHYY2016-05
Record Dates: First submitted 2017-03-12; First posted 2017-04-20 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Dysmenorrhea Primary; Pain, Menstrual
Keywords: primary dysmenorrhea; extracorporeal shock wave therapy; traditional Chinese medicine
MeSH Terms: conditions — Dysmenorrhea | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESWT during PD (Experimental): For women with primary dysmenorrhea, they have new devise Extracorporeal Shock Wave Therapy to treat. The dose is 15 hertz, 1.8-2.2bar and total 5000 frequencies approximately. The time is menstrual cycle first one and third day, and the therapy divide into two times.
  Interventions: Other: extracorporeal shock wave therapy
- ESWT before PD (Experimental): For women with primary dysmenorrhea, they have new devise Extracorporeal Shock Wave Therapy to treat. The dose is 15 hertz, 1.8-2.2 bar and total 5000 frequencies approximately. The time start from the 5th and 7th day before the estimated first day of menstrual cycle and all therapy time consuming need 15 minutes.
  Interventions: Other: extracorporeal shock wave therapy
- hot compress paste (Placebo Comparator): In hot compress paste group , the women with primary dysmenorrhea stick the hot compress paste on their belly autonomously.
  Interventions: Other: hot compress paste

INTERVENTIONS:
Other: extracorporeal shock wave therapy — Intervention group is by extracorporeal shock wave therapy.A radial shock wave device (EMS Swiss Dolor, Munich, Germany) was used. Radial shock wave is created ballistically with the pressurized air source accelerating a bullet to strike a metal applicator. The kinetic energy produced is transformed into radially expanding shock waves from the application site into the tissue to be treated. The treatment of area is lower abdomen which has some acupuncture points such as Shenque(CV8) ,Qihai(BL24), Guanyuan(CV4), Zhongji(CV3), Tianshu(ST25), Guilai(ST29) and Zigong(EX-CA1) at the right and left sides of the lower abdomen. All acupuncture points should be placed according to participants' feedback during treatment.
  Arms: ESWT before PD; ESWT during PD
Other: hot compress paste — Hot compress pastes will be sticked on the lower abdomen.
  Arms: hot compress paste

SUMMARY:
Primary dysmenorrhea (PD) is a common female disease during menstruating. Although nonsteroidal anti-inflammatory drug is an effective treatment, there are concerns about side effects. Alternative therapies, including acupuncture and moxibustion, are commonly used for PD. Nevertheless, traditional Chinese medicine takes longer period than Western medicine to release PD. Extracorporeal shock wave therapy (ESWT) originally for the treatment of musculoskeletal diseases has characteristics of fast curative effect and no wound. Currently there is no report about clinical use of ESWT for the treatment of PD. Our study is to determine whether ESWT is effective in the treatment of PD based on meridian theory of traditional Chinese medicine. The investigators hypothesis that ESWT during PD is more effective than ESWT before PD or abdominal hot paste during PD without ESWT.

DETAILED DESCRIPTION:
This randomized sham-controlled trial is to determine whether ESWT is effective in the treatment of PD. Patients are randomly divided into 3 groups: 1. ESWT treatment during PD (n=15）; 2. ESWT treatment before PD（n=15）; 3. abdominal hot paste during PD without ESWT（n=15）.

Exclusion criteria: secondary PD, concomitant chronic disease (epilepsy, gastrointestinal, cardiovascular and renal diseases), taken oral contraceptives or vitamin/ mineral supplements in the past 3 months, taking part in other clinical trials.

Medical history will be recorded before the treatment. A questionnaire will be filled by the participant. Blood samples will be collected before and after the treatment. Participants will be followed up closely by a professional nurse. Participants in group 1 will receive ESWT treatment on day1 and day 3 of each menstrual cycle. Participants in group 2 will receive twice ESWT treatment one week before the estimated first day of the menstrual cycle. Participants in group 3 will receive hot compress paste on their belly 2 inches under the navel whenever they feel painful during the menstrual cycle. Patients with PD are treated for three menstrual cycles and followed by three menstrual cycles. Evaluation time point will be one-menstrual cycle baseline, third-menstrual cycle treatment, and third-menstrual cycle follow-up period. The investigators will inform participants to keep warm, avoid cold drink and have a healthy lifestyle via telephone communication each week during the trial.

The plasma concentrations of prostaglandin F2a metabolite, PGE2, visual analogue scale (VAS), and pictorial blood loss assessment chart (PBLA), total pain relief over 4 consecutive hours (TOPAR4), Self-Rating Anxiety Scale (SAS) and other questionnaires about menstrual pain will be recorded and evaluated before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with PD ;
* women aged from 18 to 30 years;
* painful and relatively regular menstruation (duration of menstrual cycle 21 to 35 days) in recent three cycles with maximum pain intensity over 40 mm according to 10 cm visual analog scale (VAS), with primary dysmenorrhea pain features;
* willing to or already taking part in clinical trials;
* able to sign an informed consent

Exclusion Criteria:

* known lactose intolerance or chronic disease (including epilepsy, gastrointestinal, cardio-vascular or renal diseases);
* taking oral contraceptives, or regularly taking mineral or vitamin supplements in the past 3 months;
* women in pregnant women, or those with plans to get pregnant during any period of the trial;
* have experience of acupuncture

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2017-02-04 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | At baseline;1st, 2nd, 3rd, 4th, 5th, 6th menstrual cycle after randomization
  Visual analogue scale(VAS) change from baseline in menstrual pain intensity measured by VAS at 6 months.

SECONDARY OUTCOMES:
Self-Rating Anxiety Scale | At baseline;the first menstrual cycle after 3 menstrual cycles treatments;the first menstrual cycle after 3 following-up months
  Self-Rating Anxiety Scale is applied to assess the subject's anxiety and depression level.
prostaglandin F2a metabolite | At baseline(on the 2nd day of menstruation before treatment);on the 2nd day of menstruation cycle after 3 menstrual cycles treatment
  The plasma concentrations of prostaglandin F2α metabolite----Laboratory index
prostaglandin E2 metabolite | At baseline(on the 2nd day of menstruation before treatment);on the 2nd day of menstruation cycle after 3 menstrual cycles treatment
  The plasma concentrations of prostaglandin E2 metabolite----Laboratory index
pictorial blood loss assessment chart | At baseline;the first menstrual cycle after 3 menstrual cycles treatment;the first menstrual cycle after 3 following-up months
  The bleeding amount was measured using chart (PBAC).The chart (PBAC) was completed on menstruation days.

OTHER OUTCOMES:
total pain relief over 4 consecutive hours | 1st, 2nd, 3rd menstruation during treatment
  Total pain relief over 4 consecutive hours (TOPAR4) was completed on the first day of menstrual cycle during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Jian Yang, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng Y, Zhang J, Cai Y. Utility of Ultrasonography in Assessing the Effectiveness of Extracorporeal Shock Wave Therapy in Insertional Achilles Tendinopathy. Biomed Res Int. 2016;2016:2580969. doi: 10.1155/2016/2580969. Epub 2016 Nov 28. PMID 28004000
- [Background] Imamura M, Alamino S, Hsing WT, Alfieri FM, Schmitz C, Battistella LR. Radial extracorporeal shock wave therapy for disabling pain due to severe primary knee osteoarthritis. J Rehabil Med. 2017 Jan 19;49(1):54-62. doi: 10.2340/16501977-2148. PMID 27904912
- [Result] Dmitrovic R, Kunselman AR, Legro RS. Sildenafil citrate in the treatment of pain in primary dysmenorrhea: a randomized controlled trial. Hum Reprod. 2013 Nov;28(11):2958-65. doi: 10.1093/humrep/det324. Epub 2013 Aug 6. PMID 23925396
- [Result] Lefebvre G, Pinsonneault O, Antao V, Black A, Burnett M, Feldman K, Lea R, Robert M; SOGC. Primary dysmenorrhea consensus guideline. J Obstet Gynaecol Can. 2005 Dec;27(12):1117-46. doi: 10.1016/s1701-2163(16)30395-4. English, French. PMID 16524531
- [Result] Tomas-Rodriguez MI, Palazon-Bru A, Martinez-St John DRJ, Toledo-Marhuenda JV, Asensio-Garcia MDR, Gil-Guillen VF. Effectiveness of medical taping concept in primary dysmenorrhoea: a two-armed randomized trial. Sci Rep. 2015 Nov 13;5:16671. doi: 10.1038/srep16671. PMID 26564807